CLINICAL TRIAL: NCT00002673
Title: A PHASE II STUDY OF CELLULAR ADOPTIVE IMMUNOTHERAPY AS PROPHYLAXIS FOR CYTOMEGALOVIRUS DISEASE AFTER ALLOGENEIC BONE MARROW TRANSPLANTATION
Brief Title: Immunotherapy in Treating Patients Who Are Undergoing Bone Marrow or Peripheral Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Purpose: Supportive Care
Other Study IDs: 1011.01; FHCRC-1011.01; NCI-V95-0702; CDR0000064307 (Registry Identifier: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-05-21 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2010-06

CONDITIONS: Cancer
Keywords: stage IV breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent childhood rhabdomyosarcoma; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; disseminated neuroblastoma; recurrent neuroblastoma; recurrent Wilms tumor and other childhood kidney tumors; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; recurrent childhood lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; refractory chronic lymphocytic leukemia; stage III malignant testicular germ cell tumor; recurrent malignant testicular germ cell tumor; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; chronic idiopathic myelofibrosis; childhood acute promyelocytic leukemia (M3); testicular embryonal carcinoma; testicular choriocarcinoma; testicular teratoma; testicular yolk sac tumor; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and teratoma with seminoma; testicular embryonal carcinoma and yolk sac tumor; testicular embryonal carcinoma and yolk sac tumor with seminoma; testicular embryonal carcinoma and seminoma; testicular yolk sac tumor and teratoma; testicular yolk sac tumor and teratoma with seminoma; testicular choriocarcinoma and yolk sac tumor; testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and teratoma; testicular choriocarcinoma and seminoma; refractory hairy cell leukemia; recurrent/refractory childhood Hodgkin lymphoma; ovarian germ cell tumor; recurrent ovarian germ cell tumor; ovarian yolk sac tumor; ovarian embryonal carcinoma; ovarian polyembryoma; ovarian choriocarcinoma; ovarian teratoma; ovarian immature teratoma; ovarian mature teratoma; ovarian monodermal and highly specialized teratoma; stage II adult lymphoblastic lymphoma; stage II adult Burkitt lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; poor prognosis metastatic gestational trophoblastic tumor; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; infection; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; previously treated childhood rhabdomyosarcoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Carcinoma, Ovarian Epithelial; Neuroblastoma; Wilms Tumor; Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Testicular Neoplasms; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Primary Myelofibrosis; Teratoma, Testicular; Endodermal Sinus Tumor; Teratoma; Seminoma; Carcinoma, Embryonal; Leukemia, Hairy Cell; Recurrence; Teratoma, Ovarian; Burkitt Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Infections; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Therapeutics

INTERVENTIONS:
Procedure: infection prophylaxis and management

SUMMARY:
RATIONALE: White blood cells from donors who have been exposed to cytomegalovirus may be able to help prevent this infection from occurring in patients who are undergoing bone marrow or peripheral stem cell transplantation.

PURPOSE: Phase II trial to study the effectiveness of donated white blood cells to prevent cytomegalovirus infection in patients who are undergoing bone marrow or peripheral stem cell transplantation.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether adoptive immunotherapy comprising donor-derived CD8+, CMV-specific, major histocompatibility complex class I-restricted cytotoxic T-lymphocyte (CTL) clones (CD8+ CMV-specific CTL clones) and CD4+ CMV-specific T-helper (Th)-cell clones is effective in preventing CMV viremia and disease in CMV-positive patients with malignancies requiring allogeneic bone marrow or peripheral blood stem cell transplantation. II. Determine whether the transfer of CD4+ CMV-specific Th-cell clones to patients with deficient responses can reconstitute CD4+ Th-cell activity and augment adoptively transferred CD8+ CMV-specific CTL clones.

OUTLINE: Allogeneic CD8+ CMV-specific, major histocompatibility complex class I-restricted cytotoxic T-lymphocyte (CTL) clones (CD8+ CMV-specific CTL clones) and CD4+ CMV-specific T-helper (Th)-cell clones are harvested and cultured in vitro at least 2 weeks before bone marrow or peripheral blood stem cell (PBSC) transplantation. Bone marrow or PBSC are infused on day 0. Patients receive the first infusion of CD8+ CMV-specific CTL clones beginning between days 28 and 45 posttransplantation, followed 8 days later by the second infusion, followed 2 days later by the first infusion of CD4+ CMV-specific Th-cell clones. Patients who receive prednisone posttransplantation or have deficient CD8+ CTL responses (i.e., less than 50% of the response measured in the immunocompetent bone marrow donor) after the second infusion of CD8+ CMV-specific CTL clones receive a third infusion of CD8+ CMV-specific CTL clones and a second infusion of CD4+ CMV-specific Th-cell clones before day 67.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: See General Eligibility Criteria

PATIENT CHARACTERISTICS: See General Eligibility Criteria

PRIOR CONCURRENT THERAPY: See Disease Characteristics --Patients Characteristics-- Age: 12 to 60 Performance status: Not specified Hematopoietic: See Disease Characteristics Hepatic: Not specified Renal: Not specified

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 1995-06; Study Completion 2002-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stan Riddell, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States